CLINICAL TRIAL: NCT04095455
Title: The Effect Of Ultrasound-guided Modified Pectoral Nerves Block Versus Ketamine Plus Magnesium Infusion On Perioperative Analgesic Profile In Major Breast Cancer Surgeries: Randomized Controlled Study
Brief Title: The Effect Of Ultrasound-guided Modified Pectoral Nerves Block Versus Ketamine Plus Magnesium Infusion On Analgesic Profile In Breast Cancer Surgeries
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Salah Ahmed Abd Elgalil, Lecturer of Anesthesia and pain medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N10-2017
Record Dates: First submitted 2019-06-28; First posted 2019-09-19 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pectoral nerves block group (Active Comparator): modified pectoral nerves block was performed on the side of surgery
  Interventions: Procedure: pectoral nerves block group
- Ktamine plus Magnesium group (Active Comparator): Patients received 40 mg/kg of magnesium sulphate infusion in 100cc normal saline, as a bolus dose, in addition to 0.2mg/kg of ketamine as a bolus dose, 15 min before the induction of general anesthesia. This was followed by intraoperative continuous infusion of 10 mg/kg/h of magnesium sulphate combined with infusion of 0.1mg/kg/h ketamine that was started before skin incision and continued until completion of skin closure via infusion pump
  Interventions: Drug: Ketamine plus magnesium group
- Control Group (Active Comparator): Normal saline infusion with similar rate and volume to KM infusion was used as a placebo
  Interventions: Drug: Control group

INTERVENTIONS:
Procedure: pectoral nerves block group — ultrasound guided block of nerve supply of surgical site
  Arms: pectoral nerves block group
Drug: Ketamine plus magnesium group — Patients received 40 mg/kg of magnesium sulphate infusion in 100cc normal saline, as a bolus dose, in addition to 0.2mg/kg of ketamine as a bolus dose, 15 min before the induction of general anesthesia. This was followed by intraoperative continuous infusion of 10 mg/kg/h of magnesium sulphate combined with infusion of 0.1mg/kg/h ketamine that was started before skin incision and continued until completion of skin closure via infusion pump (Atom Syringe Pump S-1235).
  Arms: Ktamine plus Magnesium group
Drug: Control group — Normal saline infusion with similar rate and volume to KM infusion was used as a placebo.
  Arms: Control Group

SUMMARY:
Background: Postoperative pain is one of the greatest patient concerns following surgery. However, general anesthesia cannot provide adequate postoperative pain control and the routine use of parenteral opioids aggravates postoperative sedation, nausea, emesis, impaired oxygenation and depressed ventilation.

Hypothesis:

The investigators assume that both ultrasound guided Modified Pecs Block and combination of Ketamine and Magnesium sulphate infusion can achieve better analgesia in major breast cancer surgery in the form of reducing total amount of intraoperative fentanyl requirement and reducing postoperative morphine requirement and improvement of postoperative VAS scores both at rest and during shoulder movement so we plan this study to evaluate this assumption

DETAILED DESCRIPTION:
Surgery on the chest wall is relatively common and can be associated with significant postoperative discomfort and pain; and one of the most common surgical sites on the chest wall is the breast, with the main indication for breast surgery being breast cancer. Breast cancer has continued to be the most common cancer in females, accounting for approximately 31% of all newly detected cancer cases in the female population, worldwide. (1, 2) Thousands of patients undergo surgery in the mammary and axillary regions every year, and these procedures tend to cause significant acute pain and may develop in to cases of chronic pain in 25-60% of cases. (3) Pain can be controlled using systemic opioids which have a respiratory depressant effect and causing nausea and vomiting.

Also can be controlled using epidural catheter that can cause haemodynamic instability, so we are searching about how to devrease pain with less complications.

ELIGIBILITY:
Inclusion Criteria:

* female patients with American society of Anesthesia classification(ASA) II physical status undergoing major breast cancer surgery with axillary evacuation under general anesthesia.
* Patients' age from18 to 65 Years.
* Body mass index (BMI) are from 20 to 40 kg/m2.

Exclusion Criteria:

* Pregnant patients
* Patients having sensitivity or contraindication to test drugs or regional anesthesia.
* severe respiratory or cardiac disorders.
* history of psychological disorder.
* chronic pain .
* significant liver or renal insufficiency. .

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-11-12 (Actual); Primary Completion 2021-03-11 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
total morphine requirements | 24 hours postoperatively
  calculating the total dose of morphine consumed in postoperative analgesia

SECONDARY OUTCOMES:
fentanyl consumption | intraoperative period
  Total amount of fentanyl used by the anesthetic provider in the operating room
Visual analogue scale score | immediately after recovery and then at 1, 4, 8, 12, and 24 hours postoperatively.
  assessement of Pain intensity in the PACU using the visual analogue scale (VAS) scores, both at rest and during shoulder movement, a scale from 0 to 10. scores towards 0 is reveal good analgesia.
Sedation score | A sedation level recorded upon arrival to the PACU and at 1, 4, 8, 12, and 24 hours postoperatively.
  Sedation score assessement in Post Anesthesia Care Unit according to ramasy sedation score.(125) a scale from 1 to 6 with the preferred scores 2 or 3.
Nausea and vomiting | during the first post-operative 24 hours
  assessement of Nausea and vomiting Scores using a four-point verbal scale (127).lower scores are preferred.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Al Haram, Giza Governorate, Egypt